CLINICAL TRIAL: NCT03364140
Title: Clinical A Nation-wide Registry of Peripartum Cardiomyopathy: Clinical Status in Turkey
Brief Title: A Registry of Peripartum Cardiomyopathy in Turkey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Collaborators: Turkish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Meral Kayikcioglu, Prof Dr, Ege University
Other Study IDs: TKD-PPKM
Record Dates: First submitted 2017-08-09; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Peripartum Cardiomyopathy
Keywords: Peripartum Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Peripartum Cardiomyopathy; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripartum cardiomyopathy (PPCM) is a global disease with significant morbidity and mortality of young women. Its' etiology, epidemiology and treatment is not yet well described. This will be a retrospective, national, multicenter observational study, conducted in Turkey. It is expected that approximately 50 women with PPCM will be recorded.

DETAILED DESCRIPTION:
Peripartum cardiomyopathy (PPCM) is a global disease with significant morbidity and mortality of young women. Its' etiology, epidemiology and treatment is not yet well described. This will be a retrospective, national, multicenter observational study, conducted in centres in Turkey. It is expected that approximately 50 women with PPCM will be recorded.

The objectives of the study are:

To define the clinical status and clinical characteristics of PPCM in Turkey

To define the outcome of PPCM (short and long term)

To define the demographical and possible etiological factors

To define prognostic factors

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years of age
* Unexplained Heart Failure symptoms developed towards the end of pregnancy or in the first 6 months of postpartum period
* Ejection fraction less than 45% documented with echocardiography

Exclusion Criteria:

* Patients with any other known cardiac pathology

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female aged >18 years
Study Population: Female patients with unexplained Heart Failure symptoms developed towards the end of pregnancy or in the first 6 months of postpartum period
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-01-15 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome | 5 months after delivery
  mortality of the mother

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ural, MD, Study Director — Koc University Medical school
Locations (1):
- Koc University Medical School Cardiology Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No